CLINICAL TRIAL: NCT00363311
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Assessing the Efficacy and Safety of Dutasteride in Extending the Time to Progression of Low-Risk, Localized Prostate Cancer in Men Who Are Candidates for or Undergoing Expectant Management
Brief Title: Assessment Of Dutasteride (AVODART) In Extending The Time To Progression Of Low-Risk, Localized Prostate Cancer In Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVO105948
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms, Prostate
Keywords: Dutasteride Prostate Cancer Expectant management REDEEM
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dutasteride (Active Comparator): Dutasteride 0.5mg
  Interventions: Drug: Dutasteride
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Dutasteride — Dutasteride 0.5mg
  Arms: Dutasteride
Drug: Matching placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of dutasteride on the inhibition of low-risk, localized prostate cancer progression in men who would otherwise receive no active therapy (expectant management).

ELIGIBILITY:
Inclusion criteria:

* Must be male ≥48 and ≤82 years of age
* Have biopsy proven, low-risk, localized prostate cancer and active in expectant management not more than 14 months. [For the purposes of assessing subject eligibility a diagnostic biopsy must have included at least 10 cores, (< 4 cores positive and <50% of any one core positive) and must have been obtained within 8 months of screening]. If a saturation biopsy was performed (20 or more cores obtained) 2-3 cores are to be positive for prostate cancer and with <50% of any one core positive. Initial diagnosis of T1a/T1b obtained during a Transrectal ultrasound (TURP) is not allowed.
* Gleason score ≤6 [Gleason pattern 4 or above must not be present on any biopsy (initial or entry)]
* Clinical stage T1c-T2a
* Serum Prostate Specific Antigen (PSA) ≤11ng/mL. If the screening PSA value from the central laboratory is greater than 11ng/ml, one PSA retest is allowed through the central laboratory
* A life expectancy greater than five years.
* Able to swallow and retain oral medication
* Able and willing to participate in the full 3 years of the study
* Able to read and write (health outcomes questionnaires are self-administered), understand instructions related to study procedures and give written informed consent.

Exclusion criteria:

* Subject has ever been treated for prostate cancer with any of the following:
* Radiotherapy (external beam or brachytherapy)
* Chemotherapy
* Hormonal therapy (e.g., megestrol, medroxyprogesterone, cyproterone, diethylstilbestrol (DES)
* Oral glucocorticoids
* Gonadotropin-releasing hormone (GnRH) analogues (e.g., leuprolide, goserelin)
* Glucocorticoids, except inhaled or topical, are not permitted within 3 months prior to visit one
* Current and/or previous use of the following medications:
* Finasteride (Proscar, Propecia), or Dutasteride (GI198745, AVODART) exposure within 6 months prior to study entry are excluded.
* Any other investigational 5α-reductase inhibitors within the past 12 months.
* Anabolic steroids (subject must discontinued for 6 months prior to study entry to be eligible)
* Drugs with antiandrogenic properties within the past 6 months (e.g,. spironolactone, flutamide, bicalutamide, *cimetidine, *ketoconazole, metronidazole, progestational agents) NOTE: Use of dietary and herbal supplements (e.g., selenium, Vitamin E, saw palmetto) during the study is discouraged but not prohibited. All dietary and herbal supplement usage will be recorded in the case report form (CRF).

  *The use of cimetidine is permitted prior to study entry. The use of topical ketoconazole is permitted prior to and during the study.
* Prostate volume >80 cc
* Subject has had prior prostatic surgery including Transurethral needle ablation of the prostate (TUNA), TURP, Transurethral incision of the prostate (TUIP), laser treatment, thermotherapy, balloon dilatation, prosthesis, and ultrasound ablation within 3 months of enrolment
* Severe Benign Prostatic Hyperplasia (BPH) symptoms as manifested by International Prostate Symptom Score (IPSS) symptom score (calculated using the first 7 questions only) of ≥25 or >20 if already on alpha blocker therapy.
* Participation in any investigational or marketed drug trial within the 30 days prior to the first dose of study drug or anytime during the study period.
* Any unstable serious co-existing medical condition(s) including but not limited to myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to Screening visit; uncontrolled diabetes or peptic ulcer disease which is uncontrolled by medical management.
* Abnormal liver function test (greater than 2 times the upper limit of normal for alanine aminotransferase [ALT], aspartate aminotransferase [AST], or alkaline phosphatase [ALP]); or bilirubin >1.5 times the upper limit of normal.
* Serum creatinine >1.5 times the upper limit of normal.
* History of another malignancy within five years that could affect the diagnosis of prostate cancer.
* History or current evidence of drug or alcohol abuse within the last 12 months.
* History of any illness (including psychiatric) that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the subject.
* Known hypersensitivity to any 5α-reductase inhibitor or to any drug chemically related to dutasteride.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2006-07; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (77):
- United States (57):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Mission Hills, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, San Bernardino, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Newburgh, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Greenbelt, Maryland
  - GSK Investigational Site, Watertown, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Saint Cloud, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Marlton, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Elmont, New York
  - GSK Investigational Site, Garden City, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Orchard Park, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Springfield, Oregon
  - GSK Investigational Site, Bala-Cynwyd, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Williamsburg, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
- Canada (20):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Fredericton, New Brunswick
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Brantford, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Guelph, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Fleshner NE, Lucia MS, Egerdie B, Aaron L, Eure G, Nandy I, Black L, Rittmaster RS. Dutasteride in localised prostate cancer management: the REDEEM randomised, double-blind, placebo-controlled trial. Lancet. 2012 Mar 24;379(9821):1103-11. doi: 10.1016/S0140-6736(11)61619-X. Epub 2012 Jan 24. PMID 22277570
- [Derived] Moreira DM, Fleshner NE, Freedland SJ. Baseline Perineural Invasion is Associated with Shorter Time to Progression in Men with Prostate Cancer Undergoing Active Surveillance: Results from the REDEEM Study. J Urol. 2015 Nov;194(5):1258-63. doi: 10.1016/j.juro.2015.04.113. Epub 2015 May 16. PMID 25988518
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: AVO105948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVO105948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVO105948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVO105948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVO105948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVO105948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVO105948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A completed participant is defined as one who completed the 36-month treatment phase of the study and the 4-month safety follow-up phase.
Groups:
- Matching Placebo 0.5 mg Once Daily: Matching placebo 0.5 milligrams (mg) administered orally once daily for 156 weeks
- Dutasteride 0.5 mg Once Daily: Dutasteride 0.5 mg administered orally once daily for 156 weeks
Period: Overall Study
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Started | 155 | 147
Completed | 79 | 102
Not Completed | 76 | 45
Not completed — Adverse Event | 6 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Sponsor Terminated Study | 2 | 2
Not completed — Disease Progression | 46 | 26
Not completed — Non-Compliance | 1 | 1
Not completed — Participant Refused Biopsy | 1 | 0
Not completed — Prostate Volume/PSA Doubled | 1 | 0
Not completed — Participant Opted for Treatment | 1 | 0
Not completed — Participant Moved to Another Country | 1 | 0
Not completed — Participant Withdrew Waiting for Surgery | 0 | 1
Not completed — Withdrawn per Instructions of Monitor | 0 | 1
Not completed — Participant Moved to Louisiana | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Matching Placebo 0.5 mg Once Daily: Matching placebo 0.5 mg administered orally once daily for 156 weeks
- Total: Total of all reporting groups
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily | Total
Number analyzed (Participants) | 155 | 147 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (7.56) | 65.1 (7.13) | 65.0 (7.34)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 155 | 147 | 302
Race/Ethnicity, Customized [Number; unit: participants]
  White | 141 | 132 | 273
  African American | 12 | 8 | 20
  Asian | 1 | 4 | 5
  American Indian or Alaskan Native | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White and American Indian/Alaskan Native | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prostate Cancer (PCa) Progression [Restricted Crude Rate Analysis: Number of Participants With PCa Divided by Number of Participants in the Intent-to-Treat (ITT) Population Who Had >=1 Post-baseline Biopsy or Had a Progression
Description: PC progression (prog.) was defined as the earliest occurrence of primary therapy, also referred to as therapeutic prog., for PC (prostatectomy/radiation/hormonal therapy); or pathological prog., defined as 1 of the following: >=4 cores involved; >=50% of any 1 core involved; or a Gleason pattern of >=4 as a result of any on-study/for-cause biopsy. Primary Gleason grade is assigned to the most common tumor pattern; a second grade to the next most common tumor pattern. The two grades are added together to get a score. Gleason grade= 1-5; Gleason score=2-10; 5 and 10 indicate worst prognosis.
Time Frame: Year 1.5 and Overall (Years 0-3)
Population: ITT Population: all participants randomized to study treatment. Some participants dropped out of the study prior to meeting the primary endpoint for reasons other than disease progression or refused to have a biopsy performed.
Measure: Number; unit: participants
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 155 | 147
participants
  Year 1.5, n=144, 142 | 50 | 32
  Overall (Years 0-3), n= 155, 147 | 71 | 54
Statistical Analysis 1: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.009, Log Rank — Statistical data are for Year 1.5; Relative Risk Estimate = 0.56, 95% CI [0.36 to 0.87]
Statistical Analysis 2: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.007, Log Rank — Statistical data are for Overall (Years 0-3); Relative Risk Estimate = 0.61, 95% CI [0.43 to 0.88]

2. Secondary Outcome: Number of Participants With Therapeutic Progression
Description: Primary therapy, also referred to as therapeutic progression, for prostate cancer can be one of the following: prostatectomy, radiation, or hormonal therapy.
Time Frame: Year 1.5 and Overall (Years 0-3)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 155 | 147
participants
  Year 1.5 | 11 | 5
  Overall (Years 0-3) | 20 | 11
Statistical Analysis 1: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.13, Log Rank — Statistical data are for Year 1.5; Relative Risk Estimate = 0.46, 95% CI [0.16 to 1.31]
Statistical Analysis 2: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.053, Log Rank — Statistical data are for Overall (Years 0-3); Relative Risk Estimate = 0.48, 95% CI [0.22 to 1.03]

3. Secondary Outcome: Number of Participants With Pathologic Progression
Description: Pathological progression is defined as one of the following: >=4 cores involved; >=50% of any 1 core involved; or a Gleason pattern of >=4 as a result of any on-study/for-cause biopsy. The 2005 International Society of Urological Pathologists recommendations for Gleason scoring (GS) were used to grade tumors. A primary grade is assigned to the most common tumor pattern, and a second grade to the next most common tumor pattern. The two grades are added together to get a GS. The Gleason grade=1-5, with 5 having the worst prognosis. The Gleason score=2-10, with 10 having the worst prognosis.
Time Frame: Year 1.5 and Overall (Years 0-3)
Population: ITT Population. As the study progressed, participants dropped out of the study prior to meeting the primary endpoint for reasons other than disease progression or refused to have a biopsy performed.
Measure: Number; unit: participants
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 136 | 140
participants
  Year 1.5, n= 136, 139 | 39 | 27
  Overall (Years 0-3) n=136, 140 | 51 | 43
Statistical Analysis 1: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.031, Log Rank — Statistical data are for Year 1.5; Relative Risk Estimate = 0.59, 95% CI [0.36 to 0.96]
Statistical Analysis 2: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.079, Log Rank — Statistical data are for Overall (Years 0-3); Relative Risk Estimate = 0.70, 95% CI [0.46 to 1.05]

4. Secondary Outcome: Participants With at Least One Post-baseline Biopsy With the Indicated Prostate Cancer (PCa) Diagnosis
Description: All participants were required by protocol to undergo a transrectal ultrasound (TRUS)-guided 12-core prostate biopsy at 1.5 and 3 years or at the end of the study, if the participant discontinued the study early. Any for-cause biopsy (outside of protocol-mandated biopsies) 12 cores were obtained. If a for-cause biopsy occurred within 6 months prior to the protocol-mandated biopsy, the biopsy was counted as the protocol-mandated biopsy. All biopsies were reviewed and analyzed by a central pathologist.
Time Frame: Baseline to Month 18
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: participants
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 136 | 140
participants
  Participants with a PCa diagnosis | 111 | 111
  Participants with no PCa diagnosis | 25 | 29
Statistical Analysis 1: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.65, Fisher Exact

5. Secondary Outcome: Participants With at Least One Post-baseline Biopsy With the Indicated Prostate Cancer (PCa) Diagnosis for Their Final Biopsy
Description: All participants were required by protocol to undergo a TRUS-guided 12-core prostate biopsy at 1.5 and 3 years or at the end of the study, if the participant discontinued the study early. Any for-cause biopsy (outside of protocol-mandated biopsies) 12 cores were obtained. If a for-cause biopsy occurred within 6 months prior to the protocol-mandated biopsy, the biopsy was counted as the protocol-mandated biopsy. The final biopsy is defined as the latest post-baseline biopsy for which the results are available from the central pathology laboratory.
Time Frame: Years 0-3
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: participants
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 136 | 140
participants
  Participants with a PCa diagnosis | 105 | 90
  Participants with no PCa diagnosis | 31 | 50
Statistical Analysis 1: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.024, Fisher Exact

6. Secondary Outcome: Number of Cancer-positive Cores in a 12-core Biopsy
Description: All participants were required by protocol to undergo a TRUS-guided 12-core prostate biopsy at 1.5 and 3 years or at the end of the study, if the participant discontinued the study early. Any for-cause biopsy (outside of protocol-mandated biopsies) 12 cores were obtained. All biopsies were reviewed and analyzed by a central pathologist. . The final biopsy is defined as the latest post-baseline biopsy for which the results are available from the central pathology laboratory.
Time Frame: Baseline, Year 1.5, Year 3, Years 0-3 (Final biopsy)
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Mean (Standard Deviation); unit: cores
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 155 | 147
cores
  Baseline, n=155, 147 | 1.6 (0.74) | 1.6 (0.72)
  Year 1.5, n=87, 99 | 2.8 (1.82) | 2.2 (1.25)
  Year 3, n=52, 54 | 2.0 (1.17) | 2.0 (0.95)
  Years 0-3 (Final biopsy), n=105, 90 | 3.0 (2.03) | 2.5 (1.25)

7. Secondary Outcome: Change From Baseline in the Number of Cancer-positive Cores in a 12-core Biopsy at Years 1.5, 3, and 0-3
Description: All participants were required by protocol to undergo a TRUS-guided 12-core prostate biopsy at 1.5 and 3 years or at the end of the study, if the participant discontinued the study early. Any for-cause biopsy (outside of protocol-mandated biopsies) 12 cores were obtained. All biopsies were reviewed and analyzed by a central pathologist. Change from baseline was calculated as the number of cancer-positive cores at post-baseline biopsy minus the number of cancer-positive cores at baseline.
Time Frame: Baseline, Year 1.5, Year 3, Years 0-3 (Final biopsy)
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Mean (Standard Deviation); unit: cores
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 105 | 90
cores
  Year 1.5, n= 87, 99 | 1.1 (1.63) | 0.6 (1.36)
  Year 3, n=52, 54 | 2.0 (1.17) | 2.0 (0.95)
  Years 0-3 (Final biopsy), n=105, 90 | 3.0 (2.03) | 2.5 (1.25)

8. Secondary Outcome: Mean Percentage of Cancer-positive Cores in a 12-core Biopsy
Description: All participants were required by protocol to undergo a TRUS-guided 12-core prostate biopsy at 1.5 and 3 years or at the end of the study, if the participant discontinued the study early. Any for-cause biopsies (outside of protocol-mandated biopsies) 12 cores were obtained. All biopsies were reviewed and analyzed by a central pathologist. The sum of cancer positive cores and the sum of evaluated cores were used to compute the percentage (100* number of positive cores/number of evaluated cores).
Time Frame: Baseline, Year 1.5, Year 3, Years 0-3 (Final biopsy)
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Mean (Standard Deviation); unit: percentage of cores
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 155 | 147
percentage of cores
  Baseline, n= 155, 147 | 14.3 (7.30) | 14.5 (6.95)
  Year 1.5, n=87, 99 | 23.7 (15.76) | 19.0 (10.66)
  Year 3, n=52, 54 | 16.5 (9.71) | 17.3 (8.44)
  Years 0-3 (Final biopsy), n=105, 90 | 24.7 (15.66) | 21.7 (10.76)

9. Secondary Outcome: Change From Baseline in the Percentage of Cancer-positive Cores in a 12-core Biopsy at Years 1.5, 3, and 0-3
Description: All participants were required by protocol to undergo a TRUS-guided 12-core prostate biopsy at 1.5 and 3 years or at the end of the study, if the participant discontinued the study early. Any for-cause biopsy (outside of protocol-mandated biopsies) 12 cores were obtained. All biopsies were reviewed and analyzed by a central pathologist. (100 * number of positive cores/number of evaluated cores).
Time Frame: Baseline, Year 1.5, Year 3, Years 0-3 (Final biopsy)
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Mean (Standard Deviation); unit: percentage of cores
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 105 | 90
percentage of cores
  Year 1.5, n= 87, 99 | 8.4 (13.73) | 3.7 (11.97)
  Year 3, n=52, 54 | 4.1 (9.84) | 1.5 (10.03)
  Years 0-3 (Final biopsy), n=105, 90 | 10.0 (13.88) | 6.0 (11.40)

10. Secondary Outcome: Cumulative Length of Cancer Tumor Core
Description: All participants were required by protocol to undergo a TRUS-guided 12-core prostate biopsy at 1.5 and 3 years or at the end of the study, if the participant discontinued the study early. Any for-cause biopsy (outside of protocol-mandated biopsies) 12 cores were obtained. All biopsies were reviewed and analyzed by a central pathologist. Tumor length is calculated as the number of cores (12) * total tumor length/number of evaluated cores.
Time Frame: Baseline, Year 1.5, Year 3, Years 0-3 (Final biopsy)
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 155 | 147
millimeters
  Baseline, n= 155, 147 | 2.0 (1.86) | 2.1 (2.04)
  Year 1.5, n=87, 99 | 6.2 (5.99) | 4.8 (6.34)
  Year 3, n=52, 54 | 3.7 (3.82) | 3.8 (3.51)
  Years 0-3 (Final biopsy), n=105, 90 | 7.0 (7.02) | 6.1 (6.19)

11. Secondary Outcome: Change From Baseline in the Cumulative Length of Cancer Tumor Core at Years 1.5, 3, and 0-3
Description: All participants were required by protocol to undergo a TRUS-guided 12-core prostate biopsy at 1.5 and 3 years or at the end of the study, if the participant discontinued the study early. Any for-cause biopsy (outside of protocol-mandated biopsies) 12 cores were obtained. All biopsies were reviewed and analyzed by a central pathologist.
Time Frame: Baseline, Year 1.5, Year 3, Years 0-3 (Final biopsy)
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 105 | 90
millimeters
  Year 1.5, n= 87, 99 | 3.9 (5.71) | 2.5 (6.59)
  Year 3, n=52, 54 | 1.8 (3.94) | 1.5 (3.58)
  Years 0-3 (Final biopsy), n=105, 90 | 4.8 (6.70) | 3.8 (6.27)

12. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in Gleason Score (GS) on Repeat Biopsy at Year 1.5
Description: The 2005 International Society of Urological Pathologists recommendations for Gleason scoring were used to grade tumors. A primary grade is assigned to the most common tumor pattern (how the cancer cells look under a microscope), and a second grade to the next most common pattern. The two grades are added together to get a GS. Gleason grade range= 1-5; 5=worst prognosis. GS range=2-10; 10=worst prognosis. Improvement is defined as a decrease in GS from a baseline score of 6 (GS<=6; includes no cancer); worsening is defined as an increase in GS from a baseline score of 6 (GS >6).
Time Frame: Year 1.5
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: participants
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 81 | 100
participants
  Improvement | 6 | 21
  No change | 51 | 58
  Worsening | 24 | 21
Statistical Analysis 1: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in Gleason Score on Repeat Biopsy at Years 0-3
Description: as for outcome 12
Time Frame: Years 0-3 (Final Biopsy)
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: participants
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 136 | 140
participants
  Improvement | 31 | 50
  No cancer, GS 0 | 31 | 50
  No change | 83 | 71
  Worsening | 22 | 19
Statistical Analysis 1: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.039, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Number of Participants With the Indicated Total Gleason Score
Description: All on-study or for-cause biopsies were reviewed and analyzed by a central pathologist. The 2005 International Society of Urological Pathologists recommendations for Gleason scoring were used to grade the tumor. A primary grade is assigned to the most common tumor pattern (how the cancer cells look under a microscope), and a secondary grade to the next most common tumor pattern. The two grades are added together to get a GS. The Gleason grade ranges from 1 to 5, with 5 having the worst prognosis. The Gleason score ranges from 2 to 10, with 10 having the worst prognosis.
Time Frame: Years 0-3 (Final Biopsy)
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: participants
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 136 | 140
participants
  Missing (No Cancer) | 31 | 50
  GS 5 | 0 | 0
  GS 6 | 83 | 71
  GS 7, 3 (primary grade) + 4 (secondary grade) | 15 | 13
  GS 7, 4 (primary grade) + 3 (secondary grade) | 4 | 4
  GS 8 | 3 | 2
  GS 9-10 | 0 | 0

15. Secondary Outcome: Number of Biopsies With the Indicated Clinical Tumor Stage at Baseline
Description: All on-study or for-cause biopsies were reviewed and analyzed by a central pathologist. The 2005 International Society of Urological Pathologists recommendations for clinical tumor staging were used. T1c = tumor identified by needle biopsy (e.g., because of elevated prostate-specific antigen [PSA]); T2 = tumor confined within the prostate; T2a = tumor involves one-half of one lobe, but not both lobes of the prostate.
Time Frame: Baseline
Population: ITT Population
Measure: Number; unit: biopsies
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 155 | 147
biopsies
  T1c | 125 | 117
  T2a | 30 | 29
  T2c | 0 | 1
Statistical Analysis 1: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.80, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Number of Post-baseline Biopsies With the Indicated Change From Baseline in Clinical Stage
Description: All on-study or for-cause biopsies were reviewed and analyzed by a central pathologist. The National Comprehensive Network (NCCN), 2005 clinical practices guidelines in Oncology-prostate cancer were used for clinical tumor staging. T0: no evidence of primary tumor; T1: clinically inapparent tumor, neither palpable nor visible by imaging; T2: tumor confined within the prostate; T3: tumor extends through the prostate capsule; T4: tumor is fixed or invades adjacent structures other than seminal vesicles. A clinical stage of T0 in post-baseline biopsies has been interpreted as "No Worsening."
Time Frame: Months 0-18
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: biopsies
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 66 | 58
biopsies
  No Worsening (same/lower stage) | 53 | 53
  Worsening (higher stage) | 13 | 5
Statistical Analysis 1: Comparison: Matching Placebo 0.5 mg Once Daily vs Dutasteride 0.5 mg Once Daily; Test type: Superiority or Other; p = 0.12, Fisher Exact

17. Secondary Outcome: Prostate Volume (PV) LOCF
Description: Prostate volume was determined at baseline, at Year 1.5, and at Year 3. The anteroposterior, cephalocaudal, and transverse diameters of the prostate were obtained by transrectal ultrasound (TRUS) to calculate the prostate volume using the following formula:
  π/ 6 (anteroposterior width * cephalocaudal width * transverse width). Prostate volume calculated by pre-programmed equipment is unacceptable for the on-study prostate volume measurements.
Time Frame: Baseline and Years 1.5 and 3
Population: ITT Population. As the study progressed, participants dropped out of the study. Last observation carried forward (LOCF) was used.
Measure: Mean (Standard Deviation); unit: cubic centimeters (cc)
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 133 | 126
cubic centimeters (cc)
  Baseline, n=133, 126 | 44.2 (19.17) | 43.2 (15.32)
  Year 1.5, n=117, 117 | 43.1 (17.97) | 43.3 (15.12)
  Year 3, n=118, 118 | 43.0 (17.94) | 43.1 (15.24)

18. Secondary Outcome: Change From Baseline in Prostate Volume at Years 1.5 and 3
Description: Prostate volume was determined at baseline, Year 1.5, and Year 3. The anteroposterior, cephalocaudal, and transverse diameters of the prostate were obtained by transrectal ultrasound (TRUS) to calculate the prostate volume using the following formula:
  π/ 6 (anteroposterior width * cephalocaudal width * transverse width). Prostate volume calculated by pre-programmed equipment was unacceptable for the on-study prostate volume measurements.
Time Frame: Baseline and Years 1.5 and 3
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 118 | 118
cc
  Year 1.5, n=117, 117 | 0.7 (11.70) | -9.5 (10.51)
  Year 3, n=118, 118 | 3.3 (11.95) | -8.6 (10.89)

19. Secondary Outcome: Percent Change From Baseline in Prostate Volume at Years 1.5 and 3
Description: Prostate volume was determined at baseline, Year 1.5, and Year 3. The anteroposterior, cephalocaudal, and transverse diameters of the prostate were obtained by transrectal ultrasound (TRUS) to calculate the prostate volume using the following formula:
  π/ 6 (anteroposterior width * cephalocaudal width * transverse width). Prostate volume calculated by pre-programmed equipment is unacceptable for the on-study prostate volume measurements.
Time Frame: Baseline and Years 1.5 and 3
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 118 | 118
percent change
  Year 1.5, n=117, 117 | 3.7 (25.24) | -19.8 (26.90)
  Year 3, n=118, 118 | 7.7 (25.64) | -18.0 (27.98)

20. Secondary Outcome: Total Memorial Anxiety Scale Scores for Prostate Cancer (MAX-PC)
Description: The MAX-PC is a self-reported measure evaluating three aspects of PC-related anxiety: general anxiety related to PC/treatment, fear of recurrence, and anxiety related to PSA testing. The MAX-PC consists of 18 questions, each score ranging from 0 (least anxiety) to 3 (maximum anxiety). Total score is the sum of each question score, thus ranging from 0 to 54. A higher MAX-PC score indicates greater anxiety. At Months 18 and 36, participants were given an additional copy of the questionnaire and were asked to complete at home once they were notified of their PSA result and to send back to clinic.
Time Frame: Baseline and Month 3, 6, 12, 18, and 36
Population: ITT Population. As the study progressed, participants dropped out of the study or did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 151 | 146
points on a scale
  Baseline, n=151, 146 | 11.0 (9.28) | 11.3 (8.84)
  Month 3, n=150, 144 | 11.4 (8.80) | 11.4 (9.71)
  Month 6, n=152, 144 | 10.9 (9.01) | 10.4 (9.33)
  Month 12, n=152, 144 | 10.7 (8.82) | 9.7 (8.93)
  Month 18, n=152, 144 | 10.5 (8.96) | 9.5 (9.43)
  Month 18 Take-Home, n=152, 144 | 11.4 (9.53) | 10.6 (9.98)
  Month 36, n=152, 144 | 11.3 (9.56) | 9.6 (9.75)
  Month 36 Take-Home, n=152, 144 | 11.5 (9.68) | 9.4 (9.85)

21. Secondary Outcome: Change From Baseline in Total Memorial Anxiety Scale Scores for Prostate Cancer (MAX-PC) LOCF
Description: as for outcome 20
Time Frame: Baseline and Months 3, 6, 12, 18, and 36
Population: ITT Population. Only participants with both available baseline and post-baseline values were analyzed at the indicated time points. As the study progressed, participants dropped out of the study or did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 148 | 143
points on a scale
  Month 3, n=146, 143 | 0.4 (5.86) | 0.3 (7.04)
  Month 6, n=148, 143 | -0.0 (6.79) | -0.8 (7.15)
  Month 12, n=148, 143 | -0.1 (7.20) | -1.4 (7.58)
  Month 18, n=148, 143 | -0.3 (7.57) | -1.6 (8.25)
  Month 18 Take-Home, n=148, 143 | 0.6 (8.39) | -0.6 (8.45)
  Month 36, n=148, 143 | 0.5 (8.17) | -1.5 (8.30)
  Month 36 Take-Home, n=148, 143 | 0.7 (8.66) | -1.8 (8.22)

22. Secondary Outcome: Total MAX-PC Anxiety Subscale Score Related to PSA Testing
Description: The MAX-PC anxiety subscale consists of 3 questions related to PSA testing; "I have been so anxious about my PSA test that I have thought about delaying it.", "I have been so worried about my PSA test result that I have thought about asking my doctor to repeat the test.", "I have been so concerned about my PSA test result that I have thought about having the test repeated at another laboratory to make sure the test results were accurate." A higher MAX-PC score indicates greater anxiety.Scores range from 0 to 3 for each question. The total score is the sum of the 3 question scores; 0 to 9.
Time Frame: Baseline and Months 3, 6, 12, 18, and 36
Population: ITT Population. As the study progressed, participants dropped out of the study or did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 154 | 147
points on a scale
  Baseline, n=154, 147 | 7.1 (6.55) | 7.3 (6.35)
  Month 3, n=152, 144 | 7.5 (6.16) | 7.5 (6.95)
  Month 6, n=152, 144 | 7.0 (6.49) | 6.9 (6.60)
  Month 12, n=152, 144 | 7.0 (6.27) | 6.6 (6.46)
  Month 18, n=152, 144 | 6.7 (6.25) | 6.4 (6.78)
  Month 18 Take-Home, n=152, 144 | 7.2 (6.75) | 7.1 (7.10)
  Month 36, n=152,144 | 7.3 (6.58) | 6.5 (6.72)
  Month 36 Take-Home, n=152, 144 | 7.4 (6.64) | 6.2 (6.95)

23. Secondary Outcome: Change From Baseline in MAX-PC Anxiety Subscale Score Related to PSA Testing (LOCF)
Description: as for outcome 22
Time Frame: Baseline and Months 3, 6, 12, 18, and 36
Population: ITT Population. As the study progressed, participants dropped out of the study or did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 151 | 144
points on a scale
  Month 3 | 0.7 (4.51) | 0.3 (5.12)
  Month 6 | 0.1 (5.08) | -0.3 (5.53)
  Month 12 | 0.1 (5.28) | -0.6 (5.76)
  Month 18 | -0.2 (5.40) | -0.8 (6.08)
  Month 18 Take-Home | 0.3 (6.10) | -0.1 (6.32)
  Month 36 | 0.4 (5.80) | -0.7 (5.97)
  Month 36 Take-Home | 0.5 (5.99) | -1.0 (5.91)

24. Secondary Outcome: Total MAX-PC Fear of Recurrence Subscale Score
Description: The MAX-PC fear of recurrence subscale consists of 4 questions related to fear of recurrence; "Because cancer is unpredictable, I feel I cannot plan for the future.", "My fear of having my cancer getting worse gets in the way of my enjoying life.", "I am afraid of my cancer getting worse.", "I am more nervous since I was diagnosed with prostate cancer." A higher MAX-PC score indicates greater anxiety. Scores range from 0 to 3 for each question. The total score is the sum of the 4 question scores: 0 to 12.
Time Frame: Baseline and Months 3, 6, 12, 18, and 36
Population: ITT Population. As the study progressed, participants dropped out of the study or did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 152 | 144
points on a scale
  Baseline, n=151, 146 | 3.4 (2.51) | 3.4 (2.40)
  Month 3, n=150, 144 | 3.2 (2.59) | 3.3 (2.66)
  Month 6, n=152, 144 | 3.3 (2.57) | 2.9 (2.39)
  Month 12, n=152, 144 | 3.2 (2.51) | 2.6 (2.37)
  Month 18, n=152, 144 | 3.3 (2.52) | 2.7 (2.50)
  Month 18 Take-Home, n=152, 144 | 3.4 (2.49) | 3.0 (2.70)
  Month 36, n=152, 144 | 3.4 (2.67) | 2.7 (2.65)

25. Secondary Outcome: Change From Baseline in MAX-PC Fear of Recurrence Subscale Score (LOCF)
Description: as for outcome 24
Time Frame: Baseline and Months 3, 6, 12, 18, and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 148 | 143
points on a scale
  Month 3, n=146, 143 | -0.2 (2.07) | -0.0 (2.19)
  Month 6, n= 148, 143 | -0.2 (2.15) | -0.5 (2.13)
  Month 12, n=148, 143 | -0.1 (2.38) | -0.7 (2.24)
  Month 18, n=148, 143 | -0.1 (2.34) | -0.7 (2.31)
  Month 18 Take-Home, n=148, 143 | 0.0 (2.35) | -0.3 (2.56)
  Month 36, n=148, 143 | 0.0 (2.32) | -0.6 (2.64)
  Month 36 Take-Home, n=148, 143 | 0.0 (2.56) | -0.7 (2.55)

26. Secondary Outcome: Total Functional Assessment of Cancer Therapy Scale, Prostate Module (FACT-P) Score
Description: The FACT-P consists of a total of 39 questions. This scale is divided into five subscales: the Physical Well-Being Subscale (7 questions); the Social/Family Well-Being Subscale (7 questions); the Emotional Well-Being Subscale (6 questions); the Functional Well-Being Subscale (7 questions); and the Prostate Cancer Subscale (12 questions). The score for each of the 39 questions ranges from 0 to 4. The total FACT-P score thus ranges from 0 to156; a higher score indicates better quality of life.
Time Frame: Baseline and Months 18 and 36
Population: ITT Population. As the study progressed, participants dropped out of the study or did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 154 | 145
points on a scale
  Baseline, n=154, 145 | 129.9 (17.45) | 131.3 (15.07)
  Month 18, n=145, 140 | 126.9 (16.03) | 130.2 (16.29)
  Month 36, n=149, 140 | 126.6 (17.00) | 129.0 (16.85)

27. Secondary Outcome: Change From Baseline in Total FACT-P Score (LOCF)
Description: The FACT-P consists of a total of 39 questions. This scale is divided into five subscales: the Physical Well-Being Subscale (7 questions); the Social/Family Well-Being Subscale (7 questions); the Emotional Well-Being Subscale (6 questions); the Functional Well-Being Subscale (7 questions); and the Prostate Cancer Subscale (12 questions). The questionnaire was administered at baseline and at Months 18 and 36. The score for each of the 39 questions ranges from 0 to 4. The total FACT-P score thus ranges from 0 to156; a higher score indicates better QOL.
Time Frame: Baseline and Months 18 and 36
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 148 | 140
points on a scale
  Month 18, n=144, 140 | -4.2 (11.89) | -1.2 (14.61)
  Month 36, n=148, 140 | -3.7 (15.55) | -2.3 (15.74)

28. Secondary Outcome: Percent Change From Baseline in Total FACT-P Score (LOCF)
Description: as for outcome 27
Time Frame: Baseline and Months 18 and 36
Population: ITT Population. As the study progressed, participants dropped out of the study or did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 148 | 140
points on a scale
  Month 18, n=144, 140 | -2.8 (10.49) | -0.2 (13.44)
  Month 36, n=148, 140 | -1.8 (16.39) | -1.0 (14.16)

29. Secondary Outcome: Change From Baseline in FACT-P Physical Well-Being Subscale Score (LOCF)
Description: The FACT-P Physical Well-Being subscale is divided into 7 questions, and the participants rated the outcome over the past 7 days; "I have a lack of energy.", "I have nausea.", "Because of my physical condition, I have trouble meeting the needs of my family.", "I have pain.", "I am bothered by side effects of treatment.", "I feel ill.", "I am forced to spend time in bed." The score for each question ranges from 0 to 4; a lower score indicates better physical well-being. The total FACT-P score thus ranges from 0 to156; a higher score indicates a better quality of life.
Time Frame: Baseline and Months 18 and 36
Population: ITT Population. As the study progressed, participants dropped out of the study or did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 149 | 140
points on a scale
  Month 18, n=148, 140 | -0.4 (2.48) | -0.2 (2.28)
  Month 36, n=149, 140 | -0.3 (2.65) | -0.3 (2.58)

30. Secondary Outcome: Change From Baseline in FACT-P Social Well-Being Subscale Score (LOCF)
Description: The FACT-P Social Well-Being subscale is divided into 7 questions, and the participants rated the outcome over the past 7 days; "I feel close to my friends.", "I get emotional support from my family.", "I get support from my friends.", "My family has accepted my illness.", "I am satisfied with family communication about my illness.", "I feel close to my partner (or the person who is my main support).", "I am satisfied with my sex life." The score for each question ranges from 0 to 4; a higher score indicates better social well-being. The total FACT-P score thus ranges from 0 to 156.
Time Frame: Baseline and Months 18 and 36
Population: ITT Population. As the study progressed, participants dropped out of the study or did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Number analyzed (Participants) | 149 | 140
points on a scale
  Month 18, n=148, 140 | -1.4 (5.32) | -0.6 (5.95)
  Month 36, n=149, 140 | -1.1 (6.04) | -1.2 (6.59)

ADVERSE EVENTS:
Arm/Group | Matching Placebo 0.5 mg Once Daily | Dutasteride 0.5 mg Once Daily
Serious Adverse Events (participants affected / at risk) | 23/155 | 22/147
Other Adverse Events (participants affected / at risk) | 67/155 | 56/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo 0.5 mg Once Daily (N=155) | Dutasteride 0.5 mg Once Daily (N=147)
Coronary artery disease (Cardiac disorders) | 2 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer stage 0 with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Celulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Urospepsis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Bipoplar disorder (Psychiatric disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Cardiac pacemaker replacement (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo 0.5 mg Once Daily (N=155) | Dutasteride 0.5 mg Once Daily (N=147)
Erectile dysfunction (Reproductive system and breast disorders) | 14 | 13
Nasopharyngitis (Infections and infestations) | 15 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 13
Urinary tract infection (Infections and infestations) | 11 | 7
Fatigue (General disorders) | 9 | 7
Libido decreased (Reproductive system and breast disorders) | 6 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8
Hypertension (Vascular disorders) | 10 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Sinusitis (Infections and infestations) | 4 | 8
Pollakiuria (Renal and urinary disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.